CLINICAL TRIAL: NCT05695417
Title: A Phase 1B, Multicenter, Double-Masked, Randomized, Parallel Group Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-TKI (Axitinib Implant) for Intravitreal Injection in Subjects With Moderately Severe to Severe Non-proliferative Diabetic Retinopathy
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-TKI in Subjects With Moderately Severe to Severe Non-proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTX-TKI-2022-101
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Non-proliferative Diabetic Retinopathy
Keywords: Nonproliferative diabetic retinopathy; Diabetic retinopathy OTX-TKI
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: 2:1
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTX-TKI (Active Comparator)
  Interventions: Drug: OTX-TKI
- Sham (Sham Comparator)
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: OTX-TKI — Injection of OTX-TKI
  Arms: OTX-TKI
Drug: Sham — Sham Injection of OTX-TKI
  Arms: Sham

SUMMARY:
Evaluate the Safety, Tolerability, and Efficacy of OTX-TKI in Subjects with Moderately Severe to Severe Non-proliferative Diabetic Retinopathy

DETAILED DESCRIPTION:
Multicenter, Double-Masked, Randomized, Parallel Group Study to Evaluate the Safety, Tolerability, and Efficacy of OTX-TKI (axitinib implant) for Intravitreal Injection in Subjects with Moderately Severe to Severe Non-proliferative Diabetic Retinopathy

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age or older
* Moderately severe to severe NPDR in the study eye defined as: DRSS levels of 47 or 53 as determined by the reading center
* Diabetes type 1 or 2
* BCVA ETDRS letter score in the study eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better)

Exclusion Criteria:

* DME within 6 months involving the center of the macula in the study eye
* Presence of DME threatening the center (within 200 microns) of the macula in the study eye
* OCT CSFT of ≥320 μm in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline up to Week 52
  Frequency of treatment emergent adverse events

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score | Baseline up to Week 52
  Best Corrected Visual Acuity (BCVA) changes from baseline
Central subfield thickness changes | Baseline up to Week 52
  Central subfield thickness changes from baseline
Rescue Therapy | Baseline up to Week 52
  Proportion of subjects receiving rescue therapy
Diabetic Retinopathy Severity Scale (DRSS) changes | Baseline up to Week 52
  Diabetic Retinopathy Severity Scale (DRSS) changes from baseline

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Ocular Therapeutix Inc, Phoenix, Arizona
  - Ocular Therapeutix, Inc., Bakersfield, California
  - Ocular Therapeutix, Inc., Augusta, Georgia
  - Ocular Therapeutix, Inc., Lemont, Illinois
  - Ocular Therapeutix, Inc., Hagerstown, Maryland
  - Ocular Therapeutix, Inc., Reno, Nevada
  - Ocular Therapeutiux, Inc., Austin, Texas
  - Ocular Therapeutix Inc, Bellaire, Texas
  - Ocular Therapeutix, Inc, San Antonio, Texas
  - Ocular Therapeutix Inc., The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Undecided